CLINICAL TRIAL: NCT05620095
Title: Multicenter Registry for pAclitaxel- Coated Balloon angioplasTy in Infrapopliteal Arterial Lesions (the ACT Study)
Brief Title: Durg Coated Balloon Angioplasty in Infrapopliteal Lesions
Acronym: Act
Status: Recruiting | Type: Observational
Sponsor: Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Xuanwu Hospital, Beijing (Other); RenJi Hospital (Other); Zhejiang University (Other); First People's Hospital of Hangzhou (Other); Second Affiliated Hospital of Suzhou University (Other); Qingdao University (Other); Chengdu University of Traditional Chinese Medicine (Other); Shanghai Zhongshan Hospital (Other); Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zibo Feng, Director of Vascular Surgery, Liyuan Hospital, Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: the Act study
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-01

CONDITIONS: Arteriosclerosis; Peripheral Artery Disease; Chronic Limb Threatening Ischemia
Keywords: Drug-coated Balloon; Angioplasty; Below the knee
MeSH Terms: conditions — Arteriosclerosis; Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: drug-coated balloon — To evaluate the effectiveness and safety of drug-coated balloon angioplasty for infrapopliteal artery lesions in patients with CLTI.

SUMMARY:
This study is a multicenter observational study designed to evaluate the the effectiveness and safety of drug-coated balloon (DCB) angioplasty for below the knee arterial lesions in patients critical with Limb Threatening Ischemia (CLTI).

DETAILED DESCRIPTION:
Patients with critical limb ischemia (Rutherford category 4-5) and significant infrapopliteal lesions appropriate for angioplasty will be enrolled in this study. Subjects will be treated with the AcoArt drug coated balloon, then follow-up will be conducted at 1, 3, 6, 12 months after index procedure. Data on wound, ischemia, foot infection (WIfI) calcifications, clinical improvements, wound healing, freedom form target- lesion revascularization, patency of the target lesion and major adverse events will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Rutherford grade 4-5.
2. Patients who understand the purpose of this study, volunteer to participate in the experiment, sign informed consent and are willing to follow up.
3. Single or sequential de novo or restenotic lesions (stenosis ≥ 70% diameter reduction or occlusion) in the infrapopliteal arteries >20 mm. Lesions should not extend beyond the ankle joint.
4. Successful wire crossing of the lesion. After the pre-dilation of the ordinary balloon, the angiography showed that there was continuous blood flow.
5. At least one of the infrapopliteal arteries received a drug-coated balloon.
6. For patients with aortoiliac artery disease and femoral-popliteal artery disease, after intravascular reconstruction, blood flow can be recanalized, and there is no residual stenosis of more than 50%.
7. In patients with lower extremity arterial thrombosis, after mechanical thrombectomy, percutaneous catheter thrombolysis, and thrombus removal, patients receiving blew the knee arterial drug balloon intervention.
8. Patients who have received DCB intervention for both lower limbs can be enrolled in the group according to the intracavitary treatment time.
9. Life expectancy> 24 months.

Exclusion Criteria:

1. Blood flow was not successfully reestablished.
2. Patients with stroke, cerebral hemorrhage, gastrointestinal hemorrhage or myocardial infarction within 3 months before enrollment.
3. Patients who are known to be allergic to heparin, aspirin, other antiplatelet drugs, contrast agents, etc.
4. Patients who have participated in clinical trials of drugs or other medical devices that interfere with this clinical trial within the past 3 months.
5. Pregnant and lactating women.
6. Patients with Berg's disease.
7. Patients requiring major amputation based on preoperative evaluation of limb infection or severe ischemia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients suffered with Chronic Limb Theratening Ischemia and with significant infrapopliteal artery lesions.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Primary sustained clinical improvement at 12 months post-procedure | 12 months
  Primary sustained clinical improvement was defined as an upward shift on the Rutherford classification (Appendix) to a level of intermittent claudication without the need for repeated TLR in surviving patients without the need for unplanned amputation.
Freedom of major limb adverse events at 12 months post-procedure | 12 months
  Major limb adverse events were defined as the composite of clinically-driven target lesion revascularization (CD-TLR); unplanned, unavoidable major amputation of the index limb; and treatment caused death.

SECONDARY OUTCOMES:
Patency of the target lesions at 1 month, 3 months, 6 months and 12 months post-interventional | 1 month, 3 months, 6 months, 12 months
  Patency includes the absence of clinically driven target lesion revascularization and/or recurrent target lesion diameter stenosis ≥50% by imaging (e.g., invasive angiography or, most commonly, duplex ultrasonography).
Procedural success rate | 72 hours
  Procedural success for peripheral revascularization is defined as both technical success and absence of major adverse events (e.g., death, stroke, myocardial infarction, acute onset of limb ischemia, index bypass graft or treated segment thrombosis, and/or need for urgent/emergent vascular surgery) within 72 hours of the index procedure.
Vascular quality of life questionnaire(VascuQol) | 1 month, 3 months, 6 months, 12 months
  The VascuQol was designed as a questionnaire containing five domains: pain (4 items), symptoms (4 items), activities (8 items), social (2 items), and emotional (7 items) to evaluate Health related quality of life (HRQL). Every item has seven response options, with scores ranging from 1 to 7. A total score is the sum of all 25 item scores divided by 25.And both the total score as well as the domain scores range from 1 (worst HRQL) to 7 (best HRQL).The lower the value, the poorer the quality of life.
  1 month, 3 months, 6 months, 12 months
Wound healing rate | 1 month, 3 months, 6 months, 12 months
  Wound healing in patients with Rutherford grade 5.
Freedom from clinically-driven target lesion revascularization(CD-TLR) rate at 1 month, 3 months, 6 months, 12 months post-procedure. | 1 month, 3 months, 6 months, 12 months
  Clinically driven target lesion revascularization is defined as target lesion revascularization performed due to target lesion diameter stenosis ≥50% and either evidence of clinical or functional ischemia (e.g., recurrent/progressive life-limiting intermittent claudication, claudication unresponsive to medical therapy, CLI) or recurrence of the clinical syndrome for which the initial procedure was performed.
Major adverse events at 1 month, 3 months, 6 months, 12 months post-procedure. | 1 month, 3 months, 6 months, 12 months
  Death, unplanned major amputation of the target limb, and CD-TLR were defined as a major adverse event.
Amputation free survival rate | 1 month, 3 months, 6 months, 12 months
  Amputation free survival rate after surgery.
Primary sustained clinical improvement | 1 month, 3 months, 6 months
  Percentage of participants that experienced primary sustained clinical improvement, specified as an improvement shift in the Rutherford classification of one class in amputation free, clinically driven target lesion revascularization (TLR) free surviving subjects.
Secondary sustained clinical improvement | 1 month, 3 months, 6 months, 12 months
  Percentage of participants that experienced a secondary sustained clinical improvement, specified as an improvement shift in the Rutherford classification of one class including the need for clinically driven TLR in amputation free surviving subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Zibo Feng, Principal Investigator — Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology; Lianrui Guo, Principal Investigator — Xuanwu Hospital, Beijing
Locations (10):
- China (10):
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Zibo Feng, Wuhan, Hubei
  - the second Affiliated Hospital of Medical College of Suzhou University, Suzhou, Jiangsu
  - Qingdao Haici hospital affiliated to Qingdao University, Qingdao, Shandong
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Renji Hospital of Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan
  - Hangzhou First People's hospital of Medical College of Zhejiang University, Hangzhou, Zhejiang
  - the First Affiliated hospital of Medicine College of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No